CLINICAL TRIAL: NCT03586830
Title: A Randomized, Double-blind Placebo-controlled, Parallel-group, Multicenter, Dose-ranging Study to Evaluate the Safety and Efficacy of JNJ-64565111 in Severely Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety and Efficacy of JNJ-64565111 in Severely Obese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108488; 64565111OBE2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-06-22; First posted 2018-07-16 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Obesity and Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- JNJ-64565111 Dose Level 1 (Experimental): Participants will receive JNJ-64565111 Dose Level 1 subcutaneously (SC) once-weekly for 12-week treatment phase.
  Interventions: Drug: JNJ-64565111 Dose Level 1
- JNJ-64565111 Dose Level 2 (Experimental): Participants will receive JNJ-64565111 Dose Level 2 SC once-weekly for 12-week treatment phase.
  Interventions: Drug: JNJ-64565111 Dose Level 2
- JNJ-64565111 Dose Level 3 (Experimental): Participants will receive JNJ-64565111 Dose Level 3 SC once-weekly for 12-week treatment phase.
  Interventions: Drug: JNJ-64565111 Dose Level 3
- Placebo (Placebo Comparator): Participants will receive placebo matching to JNJ-64565111 SC once-weekly for 12-week treatment phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64565111 Dose Level 1 — Participants will receive JNJ-64565111 Dose Level 1 SC once-weekly until Week 12.
  Arms: JNJ-64565111 Dose Level 1
Drug: JNJ-64565111 Dose Level 2 — Participants will receive JNJ-64565111 Dose Level 2 SC once-weekly until Week 12.
  Arms: JNJ-64565111 Dose Level 2
Drug: JNJ-64565111 Dose Level 3 — Participants will receive JNJ-64565111 Dose Level 3 SC once-weekly until Week 12.
  Arms: JNJ-64565111 Dose Level 3
Drug: Placebo — Participants will receive matching placebo to JNJ-64565111 SC once-weekly until Week 12.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of JNJ-64565111 compared with placebo in severely obese Type 2 Diabetes Mellitus (T2DM) participants after 12 weeks of treatment on: the percentage change in body weight from baseline and safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than or equal to (>=) 35 to less than or equal to (<=) 50 kilogram per meter square (kg/m^2) at screening
* Stable weight (that is, change of <= 5 percent [%] within 12 weeks before screening based on medical or participant reported history)
* Hemoglobin A1c of >= 6.5% and <= 9.5% at screening and meets one of the inclusion criteria as: (a) on diet and exercise alone >= 12 weeks prior to screening; (b) on stable dose of single oral antihyperglycemic agent (AHA) or dual-combination oral AHAs for >= 12 weeks prior to screening
* Women must be either: (a) Postmenopausal, or (b) Permanently sterilized or otherwise be incapable of pregnancy, or (c) Heterosexually active and practicing a highly effective method of birth control, or (d) Not heterosexually active
* Willing and able to adhere to specific the prohibitions and restrictions

Exclusion Criteria:

* History of obesity with a known secondary cause (example, Cushing's disease/syndrome)
* History of Type 1 diabetes mellitus, diabetic ketoacidosis, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Fasting C-peptide less than (<) 0.7 nanogram per milliliter (ng/mL) at screening
* Fasting fingerstick glucose of >= 270 milligram per deciliter (mg/dL) (>=15 millimoles per liter [mmol/L]) on Day 1
* Ongoing, inadequately controlled thyroid disorder as assessed by the investigator's review of the participant's medical history. Participants taking thyroid hormone replacement therapy must be on stable doses for at least 6 weeks before the screening visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (27):
- United States (27):
  - Central Research Associates, Inc., Birmingham, Alabama
  - National Research Institute, Los Angeles, California
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - Sierra Clinical Research, Roseville, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Premeir Clinical Research Institute, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - CNS HealthCare, Orlando, Florida
  - Translational Research Institute for Metabolism and Diabetes, Orlando, Florida
  - Buynak Clinical Research, Valparaiso, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - M.D. Medical Research, Oxon Hill, Maryland
  - AAMRC, Flint, Michigan
  - Alas Science Clinical Research, Henderson, Nevada
  - Prestige Clinical Research, Franklin, Ohio
  - Albert J. Weisbrot and Associates, Mason, Ohio
  - Clinical Research Institute of Southern Oregon, P.C., Medford, Oregon
  - Clinical Research Associates of Central PA, LLC, Altoona, Pennsylvania
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Dallas Diabetes & Endocrine Center at Medical City, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - Permian Research Foundation, Odessa, Texas
  - Spectrum Medical, Inc, Danville, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - National Clinical Research, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 196 participants were randomized out of which 175 participants completed study.
Groups:
- Placebo: Participants self-administered the matching placebo of JNJ-64565111 subcutaneously (SC) once-weekly throughout the 12-week treatment phase or until early discontinuation of study drug.
- JNJ-64565111 5.0 mg: Participants self-administered 5.0 milligram (mg) JNJ-64565111 SC once-weekly throughout the 12-week treatment phase or until early discontinuation of study drug.
- JNJ-64565111 7.4 mg: Participants self-administered 7.4 mg JNJ-64565111 SC once-weekly throughout the 12-week treatment phase or until early discontinuation of study drug.
- JNJ-64565111 10.0 mg: Participants self-administered 10.0 mg JNJ-64565111 SC once-weekly throughout the 12-week treatment phase or until early discontinuation of study drug.
Period: Overall Study
Arm/Group | Placebo | JNJ-64565111 5.0 mg | JNJ-64565111 7.4 mg | JNJ-64565111 10.0 mg
Started | 50 | 48 | 49 | 49
Treated | 49 | 48 | 49 | 49
Completed | 48 | 42 | 41 | 44
Not Completed | 2 | 6 | 8 | 5
Not completed — Site terminated by Sponsor | 1 | 4 | 3 | 3
Not completed — Lost to Follow-up | 0 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who had received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-64565111 5.0 mg | JNJ-64565111 7.4 mg | JNJ-64565111 10.0 mg | Total
Number analyzed (Participants) | 49 | 48 | 49 | 49 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.09) | 55.1 (9.56) | 57.8 (8.97) | 56.2 (8.57) | 56.6 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 28 | 28 | 118
  Male | 19 | 16 | 21 | 21 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 14 | 15 | 51
  Not Hispanic or Latino | 39 | 36 | 35 | 34 | 144
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 10 | 13 | 17 | 52
  White | 36 | 38 | 34 | 31 | 139
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 49 | 48 | 49 | 49 | 195

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at Week 12
Description: Percent change from baseline in body weight in kilograms (kg) at Week 12 was reported.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat (mITT) analysis set included all intent-to-treat (ITT) participants who had taken at least 1 dose of study drug and had at least 1 post-baseline body weight measurement. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | JNJ-64565111 5.0 mg | JNJ-64565111 7.4 mg | JNJ-64565111 10.0 mg
Number analyzed (Participants) | 49 | 45 | 46 | 47
Percent Change | -0.70 (0.50) | -5.25 (0.57) | -6.55 (0.56) | -7.92 (0.55)
Statistical Analysis 1: Comparison: Placebo vs JNJ-64565111 5.0 mg; Test type: Superiority; p < .001, Hochberg Approach; Difference of least square (LS) means = -4.56, 95% CI 2-sided [-6.05 to -3.06], Standard Error of Mean 0.757
Statistical Analysis 2: Comparison: Placebo vs JNJ-64565111 7.4 mg; Test type: Superiority; p < .001, Hochberg Approach; Difference of LS Means = -5.85, 95% CI 2-sided [-7.34 to -4.36], Standard Error of Mean 0.755
Statistical Analysis 3: Comparison: Placebo vs JNJ-64565111 10.0 mg; Test type: Superiority; p < .001, Hochberg Approach; Difference of LS Means = -7.23, 95% CI 2-sided [-8.70 to -5.75], Standard Error of Mean 0.748

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. An TEAE is defined as an AE with an onset after the initiation study medication and before the last study medication date of the double-blind (12-Week) treatment phase plus 35 Days.
Time Frame: Up to 16 Weeks
Population: Safety analysis set included include all randomized participants who had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-64565111 5.0 mg | JNJ-64565111 7.4 mg | JNJ-64565111 10.0 mg
Number analyzed (Participants) | 49 | 48 | 49 | 49
Participants | 28 | 30 | 39 | 36

3. Secondary Outcome: Change From Baseline in Body Weight at Week 12
Description: Change from baseline in body weight at Week 12 was reported.
Time Frame: Baseline, Week 12
Population: mITT analysis set included all ITT participants who had taken at least 1 dose of study drug and had at least 1 post-baseline body weight measurement. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | JNJ-64565111 5.0 mg | JNJ-64565111 7.4 mg | JNJ-64565111 10.0 mg
Number analyzed (Participants) | 49 | 45 | 46 | 47
kg | -0.90 (0.577) | -5.92 (0.653) | -7.34 (0.648) | -9.04 (0.635)

4. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) 5 Percent (%) Weight Loss at Week 12
Description: Number of participants with >= 5 % weight loss at Week 12 was reported.
Time Frame: Week 12
Population: mITT analysis set included all ITT participants who had taken at least 1 dose of study drug and had at least 1 post-baseline body weight measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-64565111 5.0 mg | JNJ-64565111 7.4 mg | JNJ-64565111 10.0 mg
Number analyzed (Participants) | 49 | 47 | 48 | 48
Participants | 1 | 20 | 20 | 30

ADVERSE EVENTS:
Time Frame: Up to 16 Weeks
Description: Safety analysis set included include all randomized participants who had received at least one dose of study drug.
Arm/Group | Placebo | JNJ-64565111 5.0 mg | JNJ-64565111 7.4 mg | JNJ-64565111 10.0 mg
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/48 | 1/49 | 3/49
Other Adverse Events (participants affected / at risk) | 18/49 | 25/48 | 33/49 | 30/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | JNJ-64565111 5.0 mg (N=48) | JNJ-64565111 7.4 mg (N=49) | JNJ-64565111 10.0 mg (N=49)
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Incarcerated Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | JNJ-64565111 5.0 mg (N=48) | JNJ-64565111 7.4 mg (N=49) | JNJ-64565111 10.0 mg (N=49)
Abdominal Distension (Gastrointestinal disorders) | 3 | 2 | 0 | 4
Constipation (Gastrointestinal disorders) | 2 | 4 | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2 | 6
Flatulence (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 13 | 17 | 21
Vomiting (Gastrointestinal disorders) | 0 | 8 | 12 | 17
Fatigue (General disorders) | 1 | 1 | 4 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 3
Urinary Tract Infection (Infections and infestations) | 3 | 3 | 1 | 3
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 2
Amylase Increased (Investigations) | 2 | 2 | 5 | 3
Lipase Increased (Investigations) | 2 | 2 | 3 | 6
Pancreatic Enzymes Increased (Investigations) | 0 | 1 | 4 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 5 | 7 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT03586830/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT03586830/SAP_001.pdf